CLINICAL TRIAL: NCT03938155
Title: Women's Advanced Risk-assessment in Manitoba (WARM) Hearts - Examining Cardiovascular Disease Risk in Middle Aged and Older Women
Brief Title: Women's Advanced Risk-assessment in Manitoba
Acronym: WARM
Status: Recruiting | Type: Observational
Sponsor: St. Boniface Hospital (Other)
Responsible Party: Principal Investigator, Dr. Todd A Duhamel, Principal Investigator, St. Boniface Hospital
Other Study IDs: HS22576 (H2019:063)
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Cardiovascular Disease (CVD); Cardiovascular Risk Factor; Vascular Stiffness
Keywords: female; humans; aged; cardiovascular system; cardiovascular diseases; cardiovascular diseases/epidemiology; early diagnosis; frailty; frailty elderly; prospective studies; Manitoba/epidemiology; gastrointestinal microbiome; cohort studies; cause of death; risk assessment; biomarkers; risk factors; pulse wave analysis; accelerometry; exercise; physical fitness; gender; sex; women; early detection; screening program
MeSH Terms: conditions — Cardiovascular Diseases; Disease; Frailty; Motor Activity; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — This study involves the collection of blood and stool samples to:
  * characterize gut microbiota
  * analyze triglycerides, HDL/LDL cholesterol and blood glucose
  * metabolomics
  * Biomarker analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to test the ability of novel cardiovascular disease (CVD) prognostic tools to identify women at risk for future CVD. We plan to establish a cardiovascular health screening program at the St. Boniface Hospital and to test the efficacy of these tests for predicting adverse cardiovascular outcomes amongst a cohort of 1000 Manitoban women aged 55 years and older in the 5-year period after screening.

A second purpose of this project is to identify novel CVD biomarkers that may indicate a person is at risk for cardiovascular disease. Therefore, we plan to ask participants for permission to collect and store a sample of both their blood and stool for future research.

DETAILED DESCRIPTION:
Women tend to develop heart disease approximately 10-15 years later than men, with a prevalence rate similar between sexes after women turn 55 years of age. Unfortunately, women have been under represented in cardiovascular disease (CVD) research, leading to the development of screening tools that are not able to adequately identify women at risk. Current methods of CVD risk in women in the clinical setting (Framingham Risk Score) underestimate this risk as compared to men. Thus, it appears that current screening tools are not sensitive to women's cardiovascular health, which may result in a missed diagnosis of CVD risk.

Efforts to prevent CVD focus on traditional risk factors (e.g. age, sex, smoking, cholesterol and blood pressure), which do estimate 10-year risk for heart attacks. However, this approach does not determine how well the cardiovascular system is functioning for individuals. A better approach may be the addition of non-invasive procedures to detect early stages of CVD for individual patients, which are not yet available in the primary care setting.

This project builds off of Dr. Duhamel's previous work looking at novel prognostic CVD testing in women, which successfully recruited 1030 women into "The Assessment of Large and Small Artery Elasticity for the Early Detection of Cardiovascular Disease trial (see ClinicalTrials.gov Identifier: NCT02863211)" trial in a 20 month period ending May 2017. Data from that research was presented at the 2018 Canadian Women's Heart Health Summit and identified that the addition of frailty assessments to health screening has the potential to identify women with elevated CVD risk. We are taking that knowledge forward and have developed this new trial to include additional frailty measurement approaches to determine if their addition further enhances CVD risk screening.

If this new research demonstrates that the proposed CVD risk screening approach is superior to the Framingham Risk Score (FRS) at identifying individuals who have early markers of cardiovascular disease, individuals with elevated CVD risk may be empowered to participate in interventions known to restore cardiovascular health.

Trial Objectives and Purpose

The main objective of this study is to test the ability of novel CVD prognostic tools to identify women at risk for future CVD. We plan to establish a cardiovascular health screening program at the St. Boniface Hospital and to test the efficacy of these tests for predicting adverse cardiovascular outcomes amongst a cohort of 1000 Manitoban women aged 55 years and older in the 5-year period after screening.

A second purpose of this project is to identify novel CVD biomarkers that may indicate a person is at risk for cardiovascular disease. Therefore, we plan to ask participants for permission to collect and store a sample of both their blood and stool for future research.

We are recruiting exclusively women for our study for several reasons. Women are often under-represented in cardiovascular clinical trials, which is an issue because their clinical presentation and prognosis of cardiovascular disease is different, as compared to men. For example, the assortment of traditional risk factors under estimate the risk of experiencing an adverse cardiovascular event in women, as compared to men. This is an issue because the standard method to predict future adverse cardiac events utilizes the traditional risk factors. Moreover, women who suffer a heart attack are more likely to die, have a second heart attack, develop heart failure, or consequentially suffer sudden cardiac death, as compared to men. Thus, it is important to develop new strategies to increase the predictive value of cardiovascular screening methods.

Recruitment of Subjects

We will recruit by convenience sample, 1000 Manitoban women 55 years of age and older with no previous history of CVD using print, online and media advertisements around the University of Manitoba and the Winnipeg Regional Health Authority during hosted events. Potential study participants interested in participating will contact the research coordinator in person, by email, or via telephone. The research coordinator will briefly describe the study and assess potential participants for eligibility in the study. Specifically, participants will be asked via telephone if they have been previously hospitalized for ischemic heart disease, acute myocardial infarction, stroke/transient ischemic attack, percutaneous coronary intervention, coronary artery bypass surgery, congestive heart failure, or peripheral artery disease previously).

They will then be invited to attend two testing appointments: one at the Active Living Centre at the University of Manitoba and then one at the Asper Clinical Research Institute approximately one week later. Written informed consent will be obtained after describing the nature of the study before enrolment. Sufficient time will be allowed for potential participants to provide their consent. The procedures for conducting informed consent will be documented in the study records and a copy of the signed consent will be given to the participants enrolled in the study.

Trial Design

A prospective, observational clinical trial design will be utilized to determine if the use of novel CVD prognostic tools identifies individuals that are at high risk for experiencing an adverse cardiovascular event in the 5-year period after screening.

Women that respond to the advertisements will be recruited to participate in the study. Each participant will complete the WARM Hearts protocol. A blood sample (15 ml) will also be taken to measure cholesterol, blood sugar, and novel blood-based biomarkers, such as epigenetic and genetic markers of cardiovascular disease risk. Stool samples will be collected in order to characterize the gut microbiome.

We plan to utilize each individual's Personal Health Information Number (PHIN) to follow the study participants and to determine if they experienced an adverse cardiovascular outcome using the Manitoba Centre for Health Policy Population Health Research Data Repository. The repository contains anonymized information, which is linkable across files through a fictitious number assigned to the records. We have defined adverse cardiovascular outcomes as hospitalization or death due to ischemic heart disease, acute myocardial infarction, stroke, transient ischemic attack, peripheral artery disease, percutaneous coronary intervention, coronary artery bypass surgery, congestive heart failure, prescription of cardiac medication, or new onset hypertension. This information will be assessed using information from the Manitoba Centre for Health Policy Population Health Research Data Repository and will be used to compare adverse cardiovascular events with the novel CVD screening tools to determine if they predicted which individuals were at moderate to high risk of an adverse cardiovascular event over the 5-year period after screening. All participants will be asked if they are willing to participate in future research studies. If they are, they may be contacted in regard to potential participation in additional studies conducted by the Duhamel lab group.

Study Procedures

After enrolment, patients will be asked to attend two visits approximately one week apart. Each appointment visit will last approximately 90 minutes and will comprise of the following:

* Demographic information
* Medical history
* Cognitive impairment
* Body composition, as characterized by bioelectrical impedance analysis and measurement of waist circumference
* Body mass index
* Grip strength
* Gait speed
* Fried frailty phenotype (self-reported exhaustion, unintentional weight loss, and Physical activity levels)
* Physical functioning as assessed by the Senior's Fitness Test
* Heart rate variability at rest and in response to six minutes of walking, with aerobic intensity assessed by accelerometer.
* A series of self-report questionnaires to characterize:

  1. Established cardiovascular risk factors
  2. Reproductive health (menstrual history, contraception use, pregnancy history, menopause status, hormone therapy use)
  3. Daily physical activity levels
  4. Quality of life
  5. Self-esteem
  6. Gender roles, relations and identity
  7. Sleep quality
  8. Nutrition intake
  9. Self-compassion
  10. Health anxiety
  11. Depression symptoms
* Blood sampling to measure cholesterol, blood glucose, and other markers of cardiovascular disease, such as but not limited to immune cell characterization
* Non-invasive measures of arterial stiffness
* Resting blood pressure
* Blood pressure in response to 3 minutes of moderate exercise
* Objectively assessed physical activity levels as measured by an accelerometer worn for approximately one week
* Stool sample collection to characterize gut microbiome

ELIGIBILITY:
Inclusion Criteria:

* women aged 55 and older
* possess a Manitoba Personal Health Information Number

Exclusion Criteria:

Previous hospitalization or treatment for:

* Ischemic heart disease
* Acute myocardial infarction
* Stroke/Transient ischemic attack
* Percutaneous coronary intervention
* Coronary artery bypass surgery
* Congestive heart failure
* Peripheral artery disease
* Congenital heart defects
* Arrhythmia

Additional exclusion:

* Medical advice against physical activity
* Previous participant in the Assessment of Large and Small Artery Elasticity for the Early Detection of Cardiovascular Disease (NCT02863211)

Min Age: 55 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: One-thousand female participants 55 years of age or older will be recruited through a convenience sample method. Namely, we will utilize radio interviews on popular local stations to discuss the study as well as presentations at community events related to cardiovascular health. Articles will be published in a local newspaper and poster advertisements will also be placed in key locations related to the Winnipeg Regional Health Authority. Potential study participants interested in participating will contact the research coordinator in person, by email, or via telephone.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Ischemic heart disease | 5 years post-screening
  Each individual's Personal Health Information Number (PHIN) will be utilized to follow the study participants and to determine if they experienced an adverse cardiovascular outcome using the Manitoba Centre for Health Policy (MCHP) Population Health Research Data Repository. Hospital separations abstracts, medical claims and the Drug Program Information Network will be examined to provide information on hospitalizations for cardiac diseases, cardiac procedures performed, cardiac-related and other medications used, and diagnoses with cardiac diseases. Vital statistics will also provide information on cause of death to allow for mortality rate tracking. This administrative health data will be used to compare adverse cardiovascular events with the WARM Hearts protocol results to determine if this cardiovascular screening approach predicted which individuals were at moderate to high risk of an adverse cardiovascular outcome over the five-year period after screening.
Acute myocardial infarction | 5 years post-screening
  Each individual's Personal Health Information Number (PHIN) will be utilized to follow the study participants and to determine if they experienced an adverse cardiovascular outcome using the Manitoba Centre for Health Policy (MCHP) Population Health Research Data Repository. Hospital separations abstracts, medical claims and the Drug Program Information Network will be examined to provide information on hospitalizations for cardiac diseases, cardiac procedures performed, cardiac-related and other medications used, and diagnoses with cardiac diseases. Vital statistics will also provide information on cause of death to allow for mortality rate tracking. This administrative health data will be used to compare adverse cardiovascular events with the WARM Hearts protocol results to determine if this cardiovascular screening approach predicted which individuals were at moderate to high risk of an adverse cardiovascular outcome over the five-year period after screening.
Stroke | 5 years post-screening
  Each individual's Personal Health Information Number (PHIN) will be utilized to follow the study participants and to determine if they experienced an adverse cardiovascular outcome using the Manitoba Centre for Health Policy (MCHP) Population Health Research Data Repository. Hospital separations abstracts, medical claims and the Drug Program Information Network will be examined to provide information on hospitalizations for cardiac diseases, cardiac procedures performed, cardiac-related and other medications used, and diagnoses with cardiac diseases. Vital statistics will also provide information on cause of death to allow for mortality rate tracking. This administrative health data will be used to compare adverse cardiovascular events with the WARM Hearts protocol results to determine if this cardiovascular screening approach predicted which individuals were at moderate to high risk of an adverse cardiovascular outcome over the five-year period after screening.
Transient ischemic attack | 5 years post-screening
  Each individual's Personal Health Information Number (PHIN) will be utilized to follow the study participants and to determine if they experienced an adverse cardiovascular outcome using the Manitoba Centre for Health Policy (MCHP) Population Health Research Data Repository. Hospital separations abstracts, medical claims and the Drug Program Information Network will be examined to provide information on hospitalizations for cardiac diseases, cardiac procedures performed, cardiac-related and other medications used, and diagnoses with cardiac diseases. Vital statistics will also provide information on cause of death to allow for mortality rate tracking. This administrative health data will be used to compare adverse cardiovascular events with the WARM Hearts protocol results to determine if this cardiovascular screening approach predicted which individuals were at moderate to high risk of an adverse cardiovascular outcome over the five-year period after screening.
Percutaneous coronary intervention | 5 years post-screening
  Each individual's Personal Health Information Number (PHIN) will be utilized to follow the study participants and to determine if they experienced an adverse cardiovascular outcome using the Manitoba Centre for Health Policy (MCHP) Population Health Research Data Repository. Hospital separations abstracts, medical claims and the Drug Program Information Network will be examined to provide information on hospitalizations for cardiac diseases, cardiac procedures performed, cardiac-related and other medications used, and diagnoses with cardiac diseases. Vital statistics will also provide information on cause of death to allow for mortality rate tracking. This administrative health data will be used to compare adverse cardiovascular events with the WARM Hearts protocol results to determine if this cardiovascular screening approach predicted which individuals were at moderate to high risk of an adverse cardiovascular outcome over the five-year period after screening.
Coronary artery bypass surgery | 5 years post-screening
  Each individual's Personal Health Information Number (PHIN) will be utilized to follow the study participants and to determine if they experienced an adverse cardiovascular outcome using the Manitoba Centre for Health Policy (MCHP) Population Health Research Data Repository. Hospital separations abstracts, medical claims and the Drug Program Information Network will be examined to provide information on hospitalizations for cardiac diseases, cardiac procedures performed, cardiac-related and other medications used, and diagnoses with cardiac diseases. Vital statistics will also provide information on cause of death to allow for mortality rate tracking. This administrative health data will be used to compare adverse cardiovascular events with the WARM Hearts protocol results to determine if this cardiovascular screening approach predicted which individuals were at moderate to high risk of an adverse cardiovascular outcome over the five-year period after screening.
Congestive heart failure | 5 years post-screening
  Each individual's Personal Health Information Number (PHIN) will be utilized to follow the study participants and to determine if they experienced an adverse cardiovascular outcome using the Manitoba Centre for Health Policy (MCHP) Population Health Research Data Repository. Hospital separations abstracts, medical claims and the Drug Program Information Network will be examined to provide information on hospitalizations for cardiac diseases, cardiac procedures performed, cardiac-related and other medications used, and diagnoses with cardiac diseases. Vital statistics will also provide information on cause of death to allow for mortality rate tracking. This administrative health data will be used to compare adverse cardiovascular events with the WARM Hearts protocol results to determine if this cardiovascular screening approach predicted which individuals were at moderate to high risk of an adverse cardiovascular outcome over the five-year period after screening.
Future diagnosis of hypertension | 5 years post-screening
  Each individual's Personal Health Information Number (PHIN) will be utilized to follow the study participants and to determine if they experienced an adverse cardiovascular outcome using the Manitoba Centre for Health Policy (MCHP) Population Health Research Data Repository. Hospital separations abstracts, medical claims and the Drug Program Information Network will be examined to provide information on hospitalizations for cardiac diseases, cardiac procedures performed, cardiac-related and other medications used, and diagnoses with cardiac diseases. Vital statistics will also provide information on cause of death to allow for mortality rate tracking. This administrative health data will be used to compare adverse cardiovascular events with the WARM Hearts protocol results to determine if this cardiovascular screening approach predicted which individuals were at moderate to high risk of an adverse cardiovascular outcome over the five-year period after screening.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Boniface Hospital Albrechtsen Research Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
Initial WARM Hearts study data collection is expected to be complete in late 2021. Deidentified data will be available 6-months after that. Researchers wishing to access data should contact Dr. Todd Duhamel (tduhamel@sbrc.ca; orcid.org/0000-0001-8467-4800). A data dictionary will be available upon request. An itemized list of the data you are requesting with a brief proposal that outlines your justification, hypotheses, and proposed analyses will be required. Since biological samples represent a finite resource, the proposed analyses will be considered with regard to novelty, feasibility, and ethical approval. A Data Sharing Transfer Agreement or a Material Transfer Agreement must be signed and adhered to by collaborating parties and their respective institutions. Electronic data formats will be made available through the University of Manitoba Dataverse repository, following policies and procedures consistent with Tri-Council requirements.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Biological samples in the biobank will be stored for a maximum of 10 years.

REFERENCES:
- [Derived] Rose AV, Boreskie KF, Hay JL, Thompson L, Arora RC, Duhamel TA. Protocol for the WARM Hearts study: examining cardiovascular disease risk in middle-aged and older women - a prospective, observational cohort study. BMJ Open. 2021 May 25;11(5):e044227. doi: 10.1136/bmjopen-2020-044227. PMID 34035097